CLINICAL TRIAL: NCT05695950
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Orally Administered GLPG3667 Once Daily for 24 Weeks in Adult Subjects With Dermatomyositis
Brief Title: A Study Evaluating the Effects of GLPG3667 Given as Oral Treatment for up to 24 Weeks in Adults With Dermatomyositis
Acronym: GALARISSO
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLPG3667-CL-214; 2022-501097-19-00 (EU CTIS Number)
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GLPG3667 During DB + During OLE (Experimental): Participants will receive GLPG3667 dose A orally once daily for 24 weeks in the double-blind (DB) treatment period. Eligible participants will roll-over to an open-label extension (OLE) period to receive the same dose for another 24 weeks.
  Interventions: Drug: GLPG3667
- Placebo During DB + GLPG3667 During OLE (Placebo Comparator): Participants will receive placebo matching to GLPG3667 orally once daily for 24 weeks in the DB treatment period. Eligible participants will roll-over to an OLE period to receive GLPG3667 dose A orally once daily for another 24 weeks.
  Interventions: Drug: GLPG3667; Drug: Placebo

INTERVENTIONS:
Drug: GLPG3667 — GLPG3667 capsules will be administered per dose and schedule specified in the arm description.
Drug: Placebo — Placebo matching to GLPG3667 capsules will be administered per schedule specified in the arm description.
  Arms: Placebo During DB + GLPG3667 During OLE

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of orally administered GLPG3667 once daily for 24 weeks in adult participants with dermatomyositis (DM), followed by an open-label extension (OLE) period until Week 48.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant has probable or definite DM in accordance with the ACR/EULAR criteria for at least 3 months.
* Participant with DM diagnosed in the 3 years prior to screening must have undergone cancer screening (according to local standard of care or applicable guidelines) within 1 year prior to screening. Note: The evidence of cancer screening must be documented.
* Participant must present objective evidence of active disease as defined by fulfilling 1 of the criteria below (as confirmed by the sponsor):

  * DM rash as defined by modified-Cutaneous Dermatomyositis Disease Area and Severity Index Activity Score (m-CDASI-A) ≥ 6 at screening, or
  * Creatine kinase (CK) > 4x upper limit of normal (ULN) at screening, or
  * muscle biopsy evidence of active disease within 3 months prior to screening (defined as presence of active inflammation in muscle biopsy), or
  * muscle magnetic resonance imaging showing active inflammation (edema) of the proximal skeletal muscles within 3 months prior to screening, or
  * electromyography showing acute changes, such as spontaneous activity and myopathic changes not explained by other diseases within 3 months prior to screening, or
  * any other clinical evidence of active disease as confirmed by the steering committee.
* Participant has reduced muscle strength (defined as Manual Muscle Test-8 < 142/150) and at least 2 additional abnormal core set measurements out of the following 5 at screening:

  * Physician's Global Disease Activity score > 2/10 cm on the visual analog scale (VAS),
  * Patient's Global Disease Activity score > 2/10 cm on VAS,
  * extra-muscular disease activity > 2/10 cm on VAS,
  * Health Assessment Questionnaire-Disability Index score > 0.25,
  * elevated muscle enzymes (e.g. aldolase, CK, ALT, AST, and lactate dehydrogenase) with at least 1 muscle enzyme > 1.5x ULN.
* Participant previously demonstrated failure to or intolerance to first-line treatment (defined as oral corticosteroid[s] and at least 1 other immunosuppressant/ hydroxychloroquine) OR active disease despite treatment with first-line drugs. Currently, the participant is receiving maximum 3 treatments for DM (oral corticosteroid[s] and/or allowed immunosuppressant[s]/hydroxychloroquine) for at least 3 months and is on a stable dose (defined as no change in dose, type of administration, or dose regimen) for at least 4 weeks prior to screening and during screening within maximum allowed doses as specified in the study protocol. Note: Participants receiving 1 or no concomitant treatment for DM are also eligible.
* Open Label Extension : Participant must meet both of the following inclusion criteria at Visit 8 to be eligible for participation in the OLE period of the study: participant who may benefit from open-label treatment with GLPG3667, according to the investigator's judgment; participant who completed the 24-week double-blind treatment period on investigational product.

Key Exclusion Criteria:

* Participant has cancer-associated myositis (defined as myositis diagnosed within 2 years of cancer diagnosis with the exception of basal cell carcinoma, squamous cell carcinoma of the skin, or in situ uterine cervical carcinoma that has been excised and cured). Note: At least 1 year for basal cell carcinoma and squamous cell carcinoma or 5 years for in situ uterine cervical carcinoma must have passed since the excision.
* Participant has other causes of myositis (e.g. connective tissue disease) associated DM, polymyositis, juvenile DM, inclusion body myositis, or necrotizing idiopathic inflammatory myopathies (with or without rash) with the exception of overlap with secondary Sjogren's syndrome.
* Participant has permanent muscle weakness due to muscle damage (e.g. participant is wheelchair bound or has significant muscle atrophy on magnetic resonance imaging [MRI]) or a non-DM cause (drug-induced myopathy, including glucocorticoid-induced myopathy as primary cause of muscle weakness), according to investigator's judgement.
* Participant has taken any prohibited therapies within the defined washout periods before screening, and during screening as listed in the study protocol.
* Open Label Extension : Participant meeting one or more of the criteria at Visit 8 as defined in the protocol, cannot be selected for the OLE period of this clinical study. 1. Participant has total bilirubin >1.5x ULN; however, participant with an isolated increase in total bilirubin <3 x ULN due to Gilbert's Syndrome, with normal direct bilirubin, can be enrolled in the OLE period. 2. Participant has AST or ALT >1.5 x ULN (hepatic injury), or AST or ALT >=5 x ULN if judged to be of muscular origin (and confirmed by the steering committee) at Visit 7 and Visit 8.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Total improvement score [TIS] according to the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria | Week 24
  The TIS is a score derived from the evaluation of the results from 6 core set measurements (CSMs) of myositis disease activity: Physician's Global Disease Activity Assessment; Patient's Global Disease Activity Assessment; Muscle Manual Test-8 (MMT-8); Health Assessment Questionnaire-Disability Index (HAQ-DI); Enzymes (aldolase, creatine kinase (CK), alanine aminotransferase (ALT), aspartate aminotransferase (AST), and lactate dehydrogenase (LDH); and Extra-muscular disease activity. The TIS is a scale from 0 to 100 that allows for the discrimination between minimal, moderate and major responders depending on their improvement in the combined 6 CSM.

SECONDARY OUTCOMES:
Percentage of Participants With at Least Minimal Improvement According to the ACR/EULAR Criteria | Week 24
  Minimal improvement per ACR/EULAR was defined as TIS of ≥ 20 points. The TIS is a score derived from the evaluation of the results from 6 CSMs of myositis disease activity: Physician's Global Disease Activity Assessment; Patient's Global Disease Activity Assessment; MMT-8; HAQ-DI; Enzymes (aldolase, CK, ALT, AST, and LDH; and Extra-muscular disease activity. The TIS is a scale from 0 to 100 that allows for the discrimination between minimal, moderate and major responders depending on their improvement in the combined 6 CSM.
Change From Baseline in Modified-Cutaneous DM Disease Area and Severity Index Activity Score (m-CDASI-A) at Week 24 | Week 24
  The CDASI is a clinician-scored single page instrument that separately measures activity (m-CDASI-A) and damage (m-CDASI-D) in the skin of DM participants. The m-CDASI-A consists of 3 activity measures (erythema, scale, and erosion/ulceration) assessed over 15 body areas along with the activity of Gottron's papules on hands and activity of periungual changes and alopecia. m-CDASI-A ranges from 0-100. Higher scores indicate more disease activity.
Change from baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) at Week 24 | Week 24
  The HAQ-DI is a generic rather than a disease-specific instrument, comprised of 8 sections: dressing, arising, eating, walking, hygiene, reach, grip, and activities. There are 2 or 3 questions for each section. Scoring within each section is from 0 [without any difficulty] to 3 [unable to do]. For each section the score given to that section is the worst score within the section. The 8 scores of the 8 sections are summed and divided by 8.
Change from baseline in the manual muscle test (MMT-8) at Week 24 | Week 24
  MMT-8 is a set of 8 designated muscles, 7 of them being tested bilaterally (potential score 0-140). Axial (neck flexors) testing is included, so that potential maximum MMT-8 score = 150.
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs), and TEAEs Leading to Treatment Discontinuation | Baseline (Day 1) up to Week 24
Maximum Plasma Concentration (Cmax) of GLPG3667 | Week 4
Area Under the Plasma Concentration-Time Curve (AUC) of GLPG3667 | Week 4
Plasma Trough Concentration (Ctrough) at Steady State of GLPG3667 | Week 2 predose until Week 24

OTHER OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs), and TEAEs Leading to Treatment Discontinuation | Baseline (Day 1) up to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Galapagos Study Director, Study Director — Galapagos NV
Locations (54):
- United States (8):
  - HonorHealth Neurology, Scottsdale, Arizona
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - New Access Research and Medical Center, Kendall, Florida
  - Omega Research Orlando, LLC, Orlando, Florida
  - Augusta University, Augusta, Georgia
  - St. Paul Rheumatology, Eagan, Minnesota
  - Northwell Health, LLC PRIME, Lake Success, New York
  - Altoona Center for Clinical Research, P.C., Duncansville, Pennsylvania
- Argentina (5):
  - Fundacion Respirar Consultorios Médicos Dr. Doreski, Buenos Aires
  - Hospital Cordoba, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Framingham Centro Medico, La Plata
  - Instituto Medico CER, Quilmes
- UZ Leuven, Leuven, Belgium
- Chile (2):
  - Enroll SpA, Santiago
  - BioMedica Research Group Psicomedica Clinical and Research Group, Santiago
- Colombia (3):
  - Clinica de la Costa S.A.S, Barranquilla
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - Healthy Medical Center, Zipaquirá
- Croatia (2):
  - Polyclinic Bonifarm, Zagreb
  - Solmed Polyclinic, Zagreb
- Revmatologicky Ustav, Prague, Czechia
- France (3):
  - CHU de Nice Hôpital Pasteur 2 Centre de Réf des Maladies Neuromusculaires et SLA, Nice
  - Groupe Hospitalier Pitie-Salpetriere service de médecine interne et immunologie cliniqu, Paris
  - CHU Strasbourg - Hôpital Hautepierre service de rhumatologie, Strasbourg
- Germany (3):
  - Charité - Campus Charité Mitte - Klinik für Dermatologie, Venerologie und Allergologie, Berlin
  - Helios Fachklinik Vogelsang-Gommern, Gommern
  - Universitätsklinikum Tübingen - Universitäts-Hautklinik, Tübingen
- Italy (7):
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili) Medicina Interna, Brescia
  - Azienda Ospedaliero Universitaria Policlinico. PO San Marco, Catania
  - Ospedale San Raffaele U.O. di Medicina Gen. Ind. Immunologico-Clinica, Milan
  - Azienda Ospedaliero Universitaria Pisana U.O. Reumatologia Universitaria, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas U.O. Reumatologia, Rozzano
  - Ospedale San Giovanni Bosco, Torino
- Mexico (4):
  - Medical Care & Research SA de CV, Mérida
  - Centro de Investigacion Clínica GRAMEL S.C, México
  - Consultorio de Reumatologia Hospital Angeles Lindavista, México
  - Centro de Alta Especialidad en Reumatología e Investigación del Potosí S.C., San Luis Potosí City
- Poland (4):
  - Nova Reuma Domysławska i Rusiłowicz, Spółka Partnerska Lekarza Reumatologa i Fizjoterapeuty, Bialystok
  - Centrum Medyczne Plejady, Krakow
  - Zespol Poradni Specjalistycznych Reumed, Lublin
  - Klinika Ambroziak ESTEDERM, Warsaw
- Romania (3):
  - Spitalul Clinic Colentina parent, Bucharest
  - Spitalul Clinic 'Sf. Maria' Clinica de Medicina Interna si Reumatologie, Bucharest
  - Sc Medaudio-Optica SRL, Râmnicu Vâlcea
- Spain (4):
  - Hospital Universitari Vall d'Hebron Internal Medicine Dept., Barcelona
  - Hospital Clinic de Barcelona Servicio de Medicina Interna, Barcelona
  - Hospital Universitari de Bellvitge Servicio de Cardiologia, L'Hospitalet de Llobregat
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
- United Kingdom (4):
  - St. Peter´s Hospital Dept of Rheumatology, Chertsey
  - Western General Hospital Dept of Rheumatology, Edinburgh
  - King's College Hospital Dept of Rheumatology, London
  - Salford Care Organisation Dept of Rheumatology, Salford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mammoliti O, Martina S, Claes P, Coti G, Blanque R, Jagerschmidt C, Shoji K, Borgonovi M, De Vos S, Marsais F, Oste L, Quinton E, Lopez-Ramos M, Amantini D, Brys R, Jimenez JM, Galien R, van der Plas S. Discovery of GLPG3667, a Selective ATP Competitive Tyrosine Kinase 2 Inhibitor for the Treatment of Autoimmune Diseases. J Med Chem. 2024 Jun 13;67(11):8545-8568. doi: 10.1021/acs.jmedchem.4c00769. Epub 2024 May 28. PMID 38805213